CLINICAL TRIAL: NCT03954665
Title: Can Ketone Supplementation Enhance Exercise Performance?
Brief Title: Ketone Supplementation and Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113761
Record Dates: First submitted 2019-05-06; First posted 2019-05-17 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-04

CONDITIONS: Ketosis; Exercise Performance; Ketoses, Metabolic
Keywords: Ketones; Supplementation; Exercise Performance
MeSH Terms: conditions — Ketosis | interventions — Ketones; BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Testing (Active Comparator): Baseline testing for a 10km cycle time trial and a 30s Wingate cycle test.
  Interventions: Behavioral: Baseline 10 km time trial; Behavioral: Baseline 30s Wingate
- Dietary Supplement: Exogenous Ketone Salt (Experimental): Ketone salt supplementation (0.6-0.8g•kg-1•d-1) 7-days. Participants will perform two exercise performance tests (a 10km cycle time trial and a 30s Wingate cycle test on separate days) after supplementation.
  Interventions: Behavioral: 10 km time trial; Behavioral: 30s Wingate; Dietary Supplement: Ketone

INTERVENTIONS:
Behavioral: 10 km time trial — 10 km Cycling time trial test will be conducted to examine the effects of the Exogenous Ketone Salts on time
  Arms: Dietary Supplement: Exogenous Ketone Salt
Behavioral: 30s Wingate — 30s all-out test to measure peak power output
  Arms: Dietary Supplement: Exogenous Ketone Salt
Dietary Supplement: Ketone — Supplement containing exogenous ketone salts
  Arms: Dietary Supplement: Exogenous Ketone Salt
Behavioral: Baseline 10 km time trial — A baseline 10 km Cycling time trial test will be conducted
  Arms: Baseline Testing
Behavioral: Baseline 30s Wingate — A baseline 30s all-out test to measure peak power output
  Arms: Baseline Testing

SUMMARY:
The purpose of this study is to observe the effects of exogenous ketone supplements during shorter bouts of exercise testing on twenty collegiate endurance trained athletes (18-25 years of age).

DETAILED DESCRIPTION:
Some believe very high fat diets (>70% energy) can enhance exercise performance by providing additional fuel (ketones) for energy metabolism, at least for very prolonged exercise (>3-4h). Regardless, this diet is difficult to maintain so it has been suggested that ingesting ketone salts along with a normal carbohydrate (CHO) diet might be more practical. The purpose of this study is to observe the effects of ketone salt ingestion on shorter term (up to ~15 min) exercise performance. Endurance trained (≥2 year training experience; ≥7 h/week) collegiate athletes (n=20) of similar body mass (♀; 55-60kg; ♂; 75-80kg) and age 18-25y) consuming 5-6g CHO•kg-1•d-1) will be tested before and after 1 and 7d of ketone salt (Prüvit, Carrollton TX, US) supplementation (0.6-0.8g•kg-1•d-1). Participants will perform two exercise performance tests (a 10km cycle time trial and a 30s Wingate cycle test on separate days) before and after supplementation. Blood samples (glucose, lactic acid, and ketone concentration) will be taken at: baseline and following each performance test. It is hypothesized that ketone salt supplementation will increase blood ketone concentration but will not enhance these exercise performance tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female Collegiate Endurance Trained Athletes
* ≥2 year training experience; ≥7 h/week
* Ages 18-25

Exclusion Criteria:

* Smoker
* Injury that will affect exercise performance
* Sedentary Behaviour
* Currently following a High Fat diet/Ketogenic diet
* Taking Beta Blockers or Hypertension Medication
* Has Respiratory, Cardiovascular and/or Neuromuscular disease that is not cleared for exercise by a physician.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
10 km Time trial | 15-20 Minutes
  10km time trial where participants will be measured on time to completion
30s Wingate | 30 seconds
  30s Wingate all out test where participants will be measured on their peak power output

SECONDARY OUTCOMES:
Blood Ketones | 1-2 hours
  Blood Ketones will be measured using a ketone meter
Blood Glucose | 1-2 hours
  Blood Glucose will be measured using a Blood glucose meter
Blood Lactate | 1-2 hours
  Blood Lactate will be measured using a lactate meter

CONTACTS AND LOCATIONS:
Overall Officials: Peter WR Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Laboratory, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waldman HS, Basham SA, Price FG, Smith JW, Chander H, Knight AC, Krings BM, McAllister MJ. Exogenous ketone salts do not improve cognitive responses after a high-intensity exercise protocol in healthy college-aged males. Appl Physiol Nutr Metab. 2018 Jul;43(7):711-717. doi: 10.1139/apnm-2017-0724. Epub 2018 Feb 16. PMID 29451991
- [Background] O'Malley T, Myette-Cote E, Durrer C, Little JP. Nutritional ketone salts increase fat oxidation but impair high-intensity exercise performance in healthy adult males. Appl Physiol Nutr Metab. 2017 Oct;42(10):1031-1035. doi: 10.1139/apnm-2016-0641. Epub 2017 Jul 27. PMID 28750585
- [Result] Volek JS, Noakes T, Phinney SD. Rethinking fat as a fuel for endurance exercise. Eur J Sport Sci. 2015;15(1):13-20. doi: 10.1080/17461391.2014.959564. Epub 2014 Oct 2. PMID 25275931